CLINICAL TRIAL: NCT00415415
Title: Disparities in CHD in the Jackson Heart Study
Brief Title: Factors Associated With Coronary Heart Disease in African Americans in the Jackson Heart Study
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1346; 1K01HL084682-01 (NIH)
Record Dates: First submitted 2006-12-20; First posted 2006-12-22 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2006-12

CONDITIONS: Cardiovascular Diseases; Coronary Disease
Keywords: Racial Disparities; Psychosocial Risk Factors; Neighborhood Socioeconomic Status; CVD; CHD
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Coronary heart disease (CHD) is the leading cause of deaths that are related to cardiovascular disease in the United States, and Mississippi's CHD mortality rate is the highest in the nation. This study will examine data from the Jackson Heart Study to determine the effect of socioeconomic status and psychosocial factors on CHD risk in African Americans in Mississippi.

DETAILED DESCRIPTION:
CHD is a disease that is characterized by narrowing of the coronary arteries that supply blood to the heart. As a result, insufficient amounts of oxygen and nutrients reach the heart, which can cause chest pain or heart attack. Studies have shown that people's socioeconomic status is associated with their health, and that African Americans experience the highest rates of heart disease in the U.S. The Jackson Heart Study (JHS) is currently being conducted in Jackson, Mississippi, and is studying the factors that influence the development of cardiovascular disease in African American men and women. This study will examine data from the JHS to determine the effect of socioeconomic status and psychosocial factors on CHD risk in African Americans in Mississippi.

This study will recruit participants from the JHS only. Participants will report to the study site at least once for 4.5 hours for baseline measurements. Visits will include measurements of body size and blood pressure, an electrocardiogram, an echocardiogram, an ultrasound of the carotid artery, blood and urine collection, a lung function test, and interviews regarding health status and sociocultural aspects of life. Follow-up evaluations will occur 5 and 10 years after starting the study. Outcomes will include self-report and electrocardiogram-defined CHD, as well as measures of various social and psychological factors.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the Jackson Heart Study
* Diagnosis of coronary heart disease

Exclusion Criteria:

* N/A

Ages: 35 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5302
Dates: Start 2000-09; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herman Taylor, MD, Principal Investigator — Professor of Medicine - University of Mississippi Medical Center
Locations (1):
- Jackson Heart Study, Jackson, Mississippi, United States

REFERENCES:
- [Derived] Chatterjee R, Davenport CA, Svetkey LP, Batch BC, Lin PH, Ramachandran VS, Fox ER, Harman J, Yeh HC, Selvin E, Correa A, Butler K, Edelman D. Serum potassium is a predictor of incident diabetes in African Americans with normal aldosterone: the Jackson Heart Study. Am J Clin Nutr. 2017 Feb;105(2):442-449. doi: 10.3945/ajcn.116.143255. Epub 2016 Dec 14. PMID 27974310
- [Derived] Joshi PH, Khokhar AA, Massaro JM, Lirette ST, Griswold ME, Martin SS, Blaha MJ, Kulkarni KR, Correa A, D'Agostino RB Sr, Jones SR, Toth PP; Lipoprotein Investigators Collaborative (LIC) Study Group. Remnant Lipoprotein Cholesterol and Incident Coronary Heart Disease: The Jackson Heart and Framingham Offspring Cohort Studies. J Am Heart Assoc. 2016 Apr 29;5(5):e002765. doi: 10.1161/JAHA.115.002765. PMID 27130348
- [Derived] Joshi PH, Toth PP, Lirette ST, Griswold ME, Massaro JM, Martin SS, Blaha MJ, Kulkarni KR, Khokhar AA, Correa A, D'Agustino RB Sr, Jones SR; Lipoprotein Investigators Collaborative (LIC) Study Group. Association of high-density lipoprotein subclasses and incident coronary heart disease: The Jackson Heart and Framingham Offspring Cohort Studies. Eur J Prev Cardiol. 2016 Jan;23(1):41-9. doi: 10.1177/2047487314543890. Epub 2014 Jul 25. PMID 25062744